CLINICAL TRIAL: NCT02402257
Title: Dissemination of a Simulation-based Mastery Learning Curriculum for Central Venous Catheter Insertion at Veterans Affairs Hospitals: A Quantitative Study
Brief Title: Central Venous Catheter Insertion Train the Trainer
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Medical Error Reduction and Certification, Inc. (Other)
Responsible Party: Principal Investigator, Jeffrey Barsuk, Associate Professor of Medicine, Director of Simulation and Patient Safety, Northwestern University
Other Study IDs: STU00089190
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: Central Venous Catheter; Simulation-based Mastery Learning; Medical Education; Patient Outcomes; Bloodstream Infection Due to Central Venous Catheter; Pneumothorax; Inadvertent Arterial Puncture
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Traditionally-trained: Patients who undergo CVC procedures by traditionally-trained providers who have not undergone simulation-based mastery learning. This could be retrospective (before the study started) or at a site where the training was not implemented.
- CVC Train the Trainer: Patients who undergo CVC procedures by providers who have participated in simulation-based mastery learning.
  Interventions: Behavioral: CVC Train the Trainer

INTERVENTIONS:
Behavioral: CVC Train the Trainer — Trainees receive a simulation-based mastery learning intervention and train-the-trainer program on central venous catheter insertion
  Groups: CVC Train the Trainer

SUMMARY:
The investigators previously successfully implemented a central venous catheter (CVC) simulation-based mastery learning (SBML) curriculum at Northwestern University. As a result, trainee skill improved, complications, including central line associated bloodstream infections (CLABSIs) decreased and the curriculum was proven cost-effective. Therefore the Veterans Administration Medical Centers (VAMC) decided to implement this training at some of their sites as a quality improvement project. The investigators will train faculty at these locations to implement the same curriculum at their individual sites. Outcome data will be collected to evaluate the outcomes of the quality improvement (QI) project (complications, infections, skills).

DETAILED DESCRIPTION:
Beginning in 2006, Northwestern University Internal Medicine and Emergency Medicine residents completed simulation-based mastery learning in central venous catheter (CVC) insertion before clinical rotations in the Medical Intensive Care Unit (MICU). This comprehensive program in central line training used repetitive practice and simulation technology to train residents to mastery standards. This study had important patient safety implications. This program resulted in improved trainee skill and reduced CVC insertion complications, including a significant decrease in the rate of central line associated bloodstream infections (CLABSI). In addition, the investigators showed that the in CVC insertion was highly cost-effective suggesting that investment in simulation training can produce significant medical care cost savings.

This curriculum has now been successfully implemented at a few other sites. Due to the investigators' success, the VA has requested that Medical Error Reduction and Certification, Inc.(MERCI) along with Northwestern University, implements the curriculum at its sites across the county as a quality improvement project. Using a train the trainer course in CVC placement, the investigators are interested in analyzing the data that the VAMC will provide to MERCI and studying the outcomes.

Four Northwestern faculty completed a CVC insertion Master trainer curriculum. One master trainer travels to each VA facility in the program to facilitate a two-day train-the-trainer course on CVC insertion SBML. Each VA facility selects one or two "faculty champions" who complete CVC insertion SBML course and learn how to teach the curriculum on day 1 and are observed training and assessing peer healthcare providers at their institution on day 2. Course materials include standardized videos and lectures, role-playing and practice with sample learners and CVC insertion assessments. In addition to the onsite master trainer, each VA facility receives necessary training materials (standardized video lectures, data collection forms, assessment tools) and equipment (CentralLineMan simulators, ultrasound) to implement the curriculum at their institution. All participants complete pre and post testing and a course evaluation questionnaire. Quantitative outcome data on learner skills and CVC insertion quality measures are collected to measure the overall success of the project.

ELIGIBILITY:
Inclusion Criteria:

1. Previously (or prospectively) collected de-identified data on trainee skill and experience
2. Previously (or prospectively) collected de-identified data on patients in the VA ICU with CVCs
3. Previously (or prospectively) collected de-identified data on mechanical complications in the ICUs

Exclusion Criteria:

1. Data not de-identified
2. Data on pts on non-ICU units
3. Data on pts without CVCs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Trainees undergoing simulation-based mastery learning for CVC insertion
  2. De-identified patient information from patients with a CVC.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2014-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The effectiveness of simulation based mastery learning for CVC insertion on CLABSIs | 3 years
  Data from infection control on central line associated bloodstream infections will be reported for all sites each month. The investigators plan to compare the trained ICU's infection rates with other ICUs at other sites in addition to comparing the trained period versus the untrained period while trainees were rotating through the MICU.

SECONDARY OUTCOMES:
The effectiveness of simulation based mastery learning for CVC insertion on mechanical complications | 3 years
  ICUs will collect information on actual CVC insertions including complications (need for line adjustment, arterial puncture, pneumothorax). The investigators plan to compare the trained ICU's complication rates with other ICUs at other sites in addition to comparing the trained period versus the untrained period while trainees were rotating through the MICU.
The effectiveness simulation based mastery learning for CVC insertion at the learner level using simulated checklist data and trainee surveys | 2 years
  Using simulated checklist data and trainee surveys, the investigators will assess the effectiveness of our intervention at the learner level.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Barsuk, MD, MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Barsuk JH, Cohen ER, Feinglass J, McGaghie WC, Wayne DB. Use of simulation-based education to reduce catheter-related bloodstream infections. Arch Intern Med. 2009 Aug 10;169(15):1420-3. doi: 10.1001/archinternmed.2009.215. PMID 19667306
- [Background] Barsuk JH, McGaghie WC, Cohen ER, O'Leary KJ, Wayne DB. Simulation-based mastery learning reduces complications during central venous catheter insertion in a medical intensive care unit. Crit Care Med. 2009 Oct;37(10):2697-701. PMID 19885989
- [Background] Barsuk JH, McGaghie WC, Cohen ER, Balachandran JS, Wayne DB. Use of simulation-based mastery learning to improve the quality of central venous catheter placement in a medical intensive care unit. J Hosp Med. 2009 Sep;4(7):397-403. doi: 10.1002/jhm.468. PMID 19753568
- [Background] Cohen ER, Feinglass J, Barsuk JH, Barnard C, O'Donnell A, McGaghie WC, Wayne DB. Cost savings from reduced catheter-related bloodstream infection after simulation-based education for residents in a medical intensive care unit. Simul Healthc. 2010 Apr;5(2):98-102. doi: 10.1097/SIH.0b013e3181bc8304. PMID 20389233
- [Background] Barsuk JH, Cohen ER, Potts S, Demo H, Gupta S, Feinglass J, McGaghie WC, Wayne DB. Dissemination of a simulation-based mastery learning intervention reduces central line-associated bloodstream infections. BMJ Qual Saf. 2014 Sep;23(9):749-56. doi: 10.1136/bmjqs-2013-002665. Epub 2014 Mar 14. PMID 24632995